CLINICAL TRIAL: NCT06451081
Title: Building Capacity and Promoting Smoking Cessation in the Community Via "Quit to Win" Contest 2024: a Randomised Controlled Trial of a Brief Behavioural Economic Intervention
Brief Title: Brief Behavioural Economic Intervention for Smoking Cessation
Acronym: QTW2024
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Council on Smoking and Health (Other)
Responsible Party: Principal Investigator, Tzu Tsun Luk, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QTW2024
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Tobacco Smoking
Keywords: cessation; tobacco; behavioural economics; nudge; opt-out
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Opt-out+ group (Experimental): Brief cessation advice + Opt-out active referral + behavioural economics mobile messaging
  Interventions: Behavioral: Brief cessation advice; Behavioral: Opt-out active referral; Behavioral: Behavioral economic mobile messaging
- Opt-out group (Experimental): Brief cessation advice + Opt-out active referral
  Interventions: Behavioral: Brief cessation advice; Behavioral: Opt-out active referral
- Opt-in group (Active Comparator): Brief cessation advice + Opt-in active referral
  Interventions: Behavioral: Brief cessation advice; Behavioral: Opt-in active referral

INTERVENTIONS:
Behavioral: Brief cessation advice — Participants will receive brief cessation advice following the AWARD (ask, warn, advise, refer, do-it-again) model:
  A: Ask about the tobacco use status; W: Warn about the hazards of tobacco use; A: Advise the smokers to quit; R: Refer the smokers to cessation services; D: Do-it-again
Behavioral: Opt-out active referral — Participants will be automatically referred to a smoking cessation service upon joining the trial, unless they choose to opt out. Contacts of participants will be delivered to a service provider of their choice or based on their living district and preferred treatment modality
  Arms: Opt-out group; Opt-out+ group
Behavioral: Behavioral economic mobile messaging — Participants will receive behavioural economics-informed messages via mobile instant messaging for 3 months
  Arms: Opt-out+ group
Behavioral: Opt-in active referral — Participants will be offered a referral to a smoking cessation service. Contacts of participants who opt-in will be delivered to a service provider of their choice
  Arms: Opt-in group

SUMMARY:
The goal of this clinical trial is to test the effectiveness of brief behavioural economic intervention in promoting smoking cessation among smokers in the community.

DETAILED DESCRIPTION:
Smoking cessation services are free and effective but underused in Hong Kong. Active referral to smoking cessation services has consistently been found effective in promoting service use and successful quitting as a stand-alone strategy or when combined with other interventions. Participants who received active referral are introduced about the cessation services in Hong Kong and offered connection to the services of their choices. Contacts of participants who agreed to be referred are transferred to the selected cessation providers, who will subsequently contact the participants for further treatment.

The current active referral intervention uses an opt-in approach, where participants are required to actively choose to be connected to the services. By leveraging behavioural economic principles, a simple yet promising strategy to strengthen the active referral intervention is to utilize an "opt-out" approach, where participants are automatically referred to the service unless they actively decline the referral. By making referral to smoking cessation services as the default choice, the investigators aim to increase the uptake of these services and thus improve smoking cessation outcomes. Additionally, mobile messaging informed by behavioural economics principles can serve as nudges to prompt smokers to initiate quitting and utilise cessation services.

The clinical trial aims to test the effectiveness of opt-out referral, with or without behavioural economic-based mobile messaging, compared to opt-in referral, in promoting smoking cessation. The trial will be nested within the 15th "Quit to Win" Smoke-free Community Campaign organised by the Hong Kong Council on Smoking and Health.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents aged 18 years or above
2. Smoke cigarette or heated tobacco product or e-cigarette daily in the past 3 months
3. Exhaled carbon monoxide level ≥4 parts per million or a positive salivary cotinine test
4. Able to communicate in and read Chinese
5. Own a smartphone with a mobile instant messaging app installed

Exclusion Criteria:

* Participating in another smoking cessation programme or using any smoking cessation drug or nicotine replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1017 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated tobacco abstinence | 6 months after randomisation
  Verified by an exhaled carbon monoxide level of <4 parts per million and a negative salivary cotinine test

SECONDARY OUTCOMES:
Biochemically validated tobacco abstinence | 3 months after randomisation
  Verified by an exhaled carbon monoxide level of <4 parts per million and a negative salivary cotinine test
Self-reported 7-day point-prevalence tobacco abstinence | 3 months after randomisation
  Tobacco abstinence in the past 7 days
Self-reported 7-day point-prevalence tobacco abstinence | 6 months after randomisation
  Tobacco abstinence in the past 7 days
Self-reported 24-hour quit attempt | 3 months after randomisation
  Tobacco abstinence for at least 24 hours
Self-reported 24-hour quit attempt | 6 months after randomisation
  Tobacco abstinence for at least 24 hours
Self-reported use of smoking cessation service | 3 months after randomisation
  Use of any smoking cessation service during the follow-up period
Self-reported use of smoking cessation service | 6 months after randomisation
  Use of any smoking cessation service during the follow-up period

OTHER OUTCOMES:
Self-reported reduction of tobacco consumption | 3 months after randomisation
  Smoking reduction by at least half of the baseline daily number of cigarettes
Self-reported reduction of tobacco consumption | 6 months after randomisation
  Smoking reduction by at least half of the baseline daily number of cigarettes

CONTACTS AND LOCATIONS:
Overall Officials: Tzu Tsun Luk, PhD, RN, Principal Investigator — The University of Hong Kong
Locations (1):
- Community sites, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang MP, Suen YN, Li WH, Lam CO, Wu SY, Kwong AC, Lai VW, Chan SS, Lam TH. Intervention With Brief Cessation Advice Plus Active Referral for Proactively Recruited Community Smokers: A Pragmatic Cluster Randomized Clinical Trial. JAMA Intern Med. 2017 Dec 1;177(12):1790-1797. doi: 10.1001/jamainternmed.2017.5793. PMID 29059277